CLINICAL TRIAL: NCT03907605
Title: Comparison of Serum Anti-Mullerian Hormone Levels Following Uterine Artery Ligation for PPH.
Brief Title: Anti-Mullerian Hormone (AMH) is a Marker for Ovarian Reserve. There Are Many Studies About AMH Changes in Ovarian Surgery, But Little is Known for Other Surgeries. We Seek to Investigate the Hormone Variations Before and After Uterine Artey Ligation for Postpartum Hemorrage (PPH)
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: amhpph
Record Dates: First submitted 2019-04-06; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Anti-Mullerian Hormone Deficiency; Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Anti-Mullerian Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: anti- mullerian hormone — All patients belong to the same group. The blood samples will be collected at the time of surgery and 3 months after surgery from the patients who need uterine artery ligation for PPH. The blood samples will be centrifuged within 2 hours after being obtained and assessed on the same day. AMH concentrations will be measured with an enzymatically amplified two-sided immunoassay

SUMMARY:
Anti-Mullerian hormone (AMH) is a marker for ovarian reserve. There are many studies about AMH changes in ovarian surgery, but little is known for other surgeries. We seek to investigate the hormone variations before and after uterine artey ligation for postpartum hemorrage (PPH)

DETAILED DESCRIPTION:
All patients belong to the same group. The blood samples will be collected at the time of surgery and 3 months after surgery from the patients who need uterine artery ligation for PPH. The blood samples will be centrifuged within 2 hours after being obtained and assessed on the same day. AMH concentrations will be measured with an enzymatically amplified two-sided immunoassay

ELIGIBILITY:
Inclusion Criteria:

* age 18- 40 years
* no systemic or endocrine diseases
* patients who had uterine artery ligation due to PPH

Exclusion Criteria:

* Pregnancy with IVF or oosit donation
* Patients with endocrinopathy, diseases which require radiotherapy and chemotherapy etc.
* Patients with BMI >40

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients who need artery ligation for PPH during C-section.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
1- Anti-Mullerian Hormone levels variation | 3 months
  Anti-Mullerian Hormone levels before and 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes